CLINICAL TRIAL: NCT00568295
Title: A Four-Week Comparative Study Evaluating Acetaminophen Extended Release (3900 mg/Day) and Rofecoxib (12.5 mg/Day and 25 mg/Day)in the Treatment of Osteoarthritis of the Knee
Brief Title: A Four-Week Study Comparing Acetaminophen Extended Release and Rofecoxib in the Treatment of Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 99-090
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-08

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Acetaminophen; rofecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acetaminophen (Experimental): Acetaminophen Extended Release: Caplets 650 mg x 2, oral, C-112-10AP
  Interventions: Drug: acetaminophen
- Refecoxib 12.5 mg (Active Comparator): Rofecoxib: Capsules 12.5 mg, oral, C-904-1A
  Interventions: Drug: Rofecoxib
- Rofecoxib 12.5 x 2 (Active Comparator): Rofecoxib: Capsules 12.5 mg x 2, oral, C-904-1A
  Interventions: Drug: Rofecoxib

INTERVENTIONS:
Drug: acetaminophen — Acetaminophen Extended Release: Caplets 650 mg x 2, oral, C-112-10AP - Subjects were instructed to dose every eight hours according to the specified dosing schedule and to record the designated parameters in the subject diary on a daily basis throughout the course of the study until the final visit at the end of Week 4 or until discontinuation of study medication.
  Other Names: Tylenol
  Arms: Acetaminophen
Drug: Rofecoxib — Rofecoxib: Capsules 12.5 mg, oral, C-904-1A - - Subjects were instructed to dose every eight hours according to the specified dosing schedule and to record the designated parameters in the subject diary on a daily basis throughout the course of the study until the final visit at the end of Week 4 or until discontinuation of study medication.
  Other Names: Viox
  Arms: Refecoxib 12.5 mg
Drug: Rofecoxib — Rofecoxib: Capsules 12.5 mg x 2, oral, C-904-1A - Subjects were instructed to dose every eight hours according to the specified dosing schedule and to record the designated parameters in the subject diary on a daily basis throughout the course of the study until the final visit at the end of Week 4 or until discontinuation of study medication.
  Other Names: Viox
  Arms: Rofecoxib 12.5 x 2

SUMMARY:
To compare acetaminophen (Tylenol) with rofecoxib (Viox) for the treatment of Osteoarthritis of the Knee

DETAILED DESCRIPTION:
An initial screening visit was performed in order to assess subject medical history and the potential eligibility of subjects. Following the initial screening visit, all potential subjects underwent a washout period from their usual arthritis medication and returned to the study center for a baseline visit to verify their eligibility.

At the completion of the baseline visit, all eligible subjects were randomly assigned to a treatment group and instructed on the dosing regimen for their assigned study medication.

Subjects returned to the study center for follow-up visits after Week 1 and Week 2 of treatment and a final visit after Week 4 of treatment or upon discontinuation from the study.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic idiopathic osteoarthritis of the knee for a minimum of six months duration requiring treatment with either an analgesic or anti-inflammatory agent on a regular basis (greater than or equal to three days/week) for at least three months.
* A history of osteoarthritis of the knee characterized by pain of at least a moderate intensity.
* Demonstrated radiographic evidence of mild to moderate osteoarthritis based on the Kellgren and Lawrence radiographic entry criteria of grade 2 or 3 osteoarthritis.
* Subjects' physical ability was to be either American College of Rheumatology (ACR) Function Class I or II
* At the baseline visit, subjects must have reported a maximum pain intensity experienced over the previous 24 hours of at least moderate on a five-point scale of none(0), mild(1), moderate(2), moderately severe(3), or severe(4) in order to be enrolled in the study.

Exclusion Criteria:

* Medical history, physical examinations, or radiographs suggestive of other types of arthritis, pseudogout, collagen vascular disease or fibromyalgia.
* Medical or psychiatric conditions that may influence absorption, metabolism, or excretion of the study medications or interfere with interpretation of adverse reactions to the study drug.
* History of allergy, sensitivity, contraindication or non-response to acetaminophen, rofecoxib, or drugs classified as NSAIDs including aspirin.
* Use of concomitant medications that might interfere with study drug assessments, including intra-articular corticosteroids.
* Signs of active knee inflammation, morning stiffness of greater than 30 minutes duration.
* Rheumatoid factor quantitative value greater than or equal to 40 IU/mL or a Westergren erythrocyte sedimentation rate greater than or equal to 40 mm/hour.
* ACR functional class III or IV, or unable to walk without assistive devices.
* Pregnancy, lactation, or expect to become pregnant within one month of study completion.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 1999-10; Primary Completion 2000-10 (Actual); Study Completion 2000-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Western Ontario and McMaster Universities (WOMAC) pain subscale score at week 4 in the per protocol study population. | Four Weeks

SECONDARY OUTCOMES:
Change from Baseline in the WOMAC pain subscale score | Weeks 1 and 2
Change from baseline in the WOMAC stiffness and physical function subscale scores | Weeks 1, 2 and 4
Investigator's impression of therapeutic response | Weeks 1, 2, and 4
Subject's assessment of medication as an analgesic for the study knee joint | Weeks 1, 2, and 4
Daily pain intensity differences from baseline | Week 1
Investigator's global impression of therapeutic response | Week 4
Subject's overall impression of the study medication | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Kuffner, MD, Study Director — McNeil Consumer Healthcare USA